CLINICAL TRIAL: NCT00656695
Title: The Comparison Between Clinical and Paraclinical Effect of Iminoral Vs Neoral in Prevention of Acute Rejection in the First Year Afer Transplantation in De Novo Renal Transplant Patients
Brief Title: Comparisone of Iminoral Versus Neoral in Prevention of Acute Rejection in Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imam Khomeini Hospital (Other)
Responsible Party: Principal Investigator, Mohammad Reza Khatami, Associate professor, Imam Khomeini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iminoral
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: End Stage Renal Disease; Renal Transplantation
Keywords: Iminoral; Neoral; Acute renal transplant rejection
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Iminoral; Cyclosporine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): taking Iminoral
  Interventions: Drug: Iminoral
- 2 (Active Comparator): taking Neoral
  Interventions: Drug: Neoral

INTERVENTIONS:
Drug: Iminoral — Iminoral in form of capsules 25,50 and 100 mg giving in the dose of 3-7 mg/kg twice daily
  Arms: 1
Drug: Neoral — Neoral in form of capsules 25,50 and 100 mg giving in the dose of 3-7 mg/kg twice daily
  Arms: 2

SUMMARY:
Cyclosporine is the key drug in organ transplantation. In Iran the investigators have more than 2500 new renal transplantation each year and because of this the government pay a huge amount of money for subsiding the imported cyclosporine in the form of Neoral. Recently an Iranian drug company introduced this drug in the name of Iminoral which has been approved by different authorities in Iran and abroad, (including the Ministry of Health in Iran and also European Directorate for the Quality of Medicines Certification Unit and FDA(Department of Health and Human Services,Center for Drug Evaluation and Research)). The investigators study is the first clinical trial to compare the effect of Iminoral versus Neoral in preventing acute rejection in renal transplantation and also to compare the side effects of these two drugs.

ELIGIBILITY:
Inclusion Criteria:

1. renal transplantation candidates
2. written consent
3. not taking participate in any other clinical trial in last 3 months

Exclusion Criteria:

1. primary FSGS
2. hyperoxaluria
3. age under 18
4. multi organ transplantation
5. any malignancy in 5 years
6. PRA > 25%
7. use of Tacrolimus
8. hyper acute rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
transplanted kidney acute rejection | one year

SECONDARY OUTCOMES:
cyclosporine side effects | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad R Khatami, MD, Principal Investigator — Imam Khomeini Hospital
Locations (1):
- Imam Khomeini Hospital, Tehran, Iran

REFERENCES:
- [Derived] Khatami SM, Taheri S, Azmandian J, Sagheb MM, Nazemian F, Razeghi E, Shahidi S, Sadri F, Shamshiri AR, Sayyah M. One-Year Multicenter Double-Blind Randomized Clinical Trial on the Efficacy and Safety of Generic Cyclosporine (Iminoral) in De Novo Kidney Transplant Recipients. Exp Clin Transplant. 2015 Jun;13(3):233-8. PMID 26086833